CLINICAL TRIAL: NCT02564601
Title: The Impact of Piano Training on Cognitive Performance and Psychosocial Well-Being in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Jennifer Bugos, Assistant Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19415
Record Dates: First submitted 2015-09-16; First posted 2015-10-01 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Aging
Keywords: intervention; cognition; aging; piano training; computer brain training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A1 Piano Training (Experimental): 16 weekly classes will be provided to the piano training group. Each piano class session will focus upon review of materials (15-20 min), and the remaining portion of the class will focus upon learning new skills and concepts. This course includes finger dexterity exercises, basic piano technique, and basic piano repertoire.
  Interventions: Behavioral: Piano Training
- A2 Computer Cognitive Training (Experimental): 16 weekly classes will be provided to the computerized cognitive training group. Computerized cognitive training involves process-based computerized practice of adaptive perceptual exercises. Each computer cognitive training class session will focus upon practice of cognitive exercises that vary in difficulty ranging from basic auditory processing speed to application through memory and working memory exercises. Within each exercise, the stimuli (i.e., tones, speech sounds, words, sentences) become less discriminable and speed of presentation increases (making the exercises more difficult) as performance improves.
  Interventions: Behavioral: Computer Cognitive Training
- A 3 No Treatment Controls (No Intervention): No classes will be provided to our control group. This is a no-treatment control group.

INTERVENTIONS:
Behavioral: Piano Training — The intervention focuses upon progressively difficult piano performance exercises (repertoire), technique, and finger dexterity exercises.
  Arms: A1 Piano Training
Behavioral: Computer Cognitive Training — The intervention focuses upon progressively difficult perceptual exercises using the Brain Fitness program plus working memory exercises.
  Arms: A2 Computer Cognitive Training

SUMMARY:
This project evaluates the effects of piano training and computerized cognitive training on cognitive performance in healthy older adults compared to controls. The project is intended for healthy older adults (60-80 years) with little to no previous musical training (less than three years of prior musical training or cognitive training and not currently engaged in music reading or musical performance, less than 10 hours of previous cognitive training). Investigators anticipate that musical engagement will serve as an enjoyable cognitive intervention for older adults. Investigators believe that piano training will enhance cognitive performance on executive functions essential for maintaining independence in older adulthood. Learning a musical instrument, while challenging, will improve self-efficacy, mood, and qualtiy of life. Participants engaged in piano training will demonstrate reduced cortisol levels and increased immune function responses. Investigators predict that adults enrolled in computerized cognitive training will demonstrate enhanced memory, working memory and self-efficacy post-training.

DETAILED DESCRIPTION:
The project purpose is to scientifically examine the benefits of piano training as compared to computer cognitive training and no treatment controls on cognitive (processing speed, task-switching, verbal fluency, verbal memory, and working memory), psychosocial (mood, self-efficacy, and quality of life), and physiological variables (biomarkers) in healthy older adult participants in a randomized clinical trial design.

Participants: Ninety community dwelling older adults will be recruited from the community. Criteria for enrollment are: between the ages of 60-80, native English speakers, not currently taking medications affecting memory performance, have no pre-existing cognitive impairment or neurological disorders, (as indicated by the Telephone Interview for Cognitive Status > 30), no moderate to severe depression (as indicated by the Geriatric Depression Scale), no difficulty with hand movements, less than three years of prior musical training, not currently engaged in music reading or musical performance, and less than ten hours of prior computer brain training experience. Participants will be randomly assigned to one of three groups stratified by intelligence and gender: piano instruction, computerized cognitive training or a no treatment control group. Informed written consent will be obtained in accordance with the Institutional Review Board.

Procedure: Participants will be tested in three visits: pre-training, immediately post-training, and three months follow-up. Those randomized to piano training or computerized cognitive training will complete their assigned training between pre-training and post-training visits. Measures of music aptitude and intelligence will be administered at the pre-training visit. These factors can influence cognitive performance. Any significant differences at baseline between the three assigned groups will be statistically controlled for in the analyses. Standardized cognitive measures will be used to examine processing speed, task-switching, verbal fluency, verbal memory, and working memory at each visit. Psychosocial outcomes (mood, self-efficacy, and quality of life) and physiological biomarkers will also be evaluated at each visit.

The goal for both interventions will be to complete 48 hours of group training over a four month period (16 weeks). Sixty participants (30 piano training; 30 auditory computer training) will be asked to attend three hours of training each week. Thirty participants will serve in the no treatment control group. Piano training will consist of basic piano technique, dexterity exercises, piano literature, and music theory. Participants will be expected to perform all major scales, repertoire from the Alfred All-in-One Method, and complete weekly theory assignments. Each class session is structured as a cognitive intervention that focuses upon review of materials (15-20 min), and the remaining portion of the class focuses upon learning new skills and concepts. Computerized cognitive training involves computerized perceptual practice exercises that vary in difficulty ranging from basic auditory processing speed to application through memory exercises. Within each exercise, the stimuli (i.e., tones, speech sounds, words, sentences) become less discriminable and speed of presentation increases (making the exercises more difficult) as performance improves. The Brain Fitness training program with working memory exercises will be used.

Data source(s). Data will consist of a series of standardized cognitive, psychosocial, and neurophysiological measures administered at three time points: pre-training, post-training, and at a three month follow-up. All standardized measures have been previously used to assess the efficacy of cognitive training approaches and demonstrate good psychometric properties.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 60-80
* native English speakers
* no pre-existing cognitive impairment or neurological impairment
* not taking medications affecting memory performance (sleep meds, antidepressants, etc.)
* Telephone Interview for Cognitive Status (score >30)
* no moderate to severe depression
* no difficulty with hand movements
* less than three years of formal music training
* no difficulty with the movement of their hands
* not currently engaged in music reading or musical performance
* < 10 hours of previous cognitive training

Exclusion Criteria:

* Those not between 60-80
* those taking medications affecting memory performance
* Non-Native English Speakers
* Those with pre-existing cognitive impairment
* Telephone Interview for Cognitive Status (score < 30)
* Those with difficulty in the movement of their hands
* Those with more than three years of formal music training or currently engaged in music reading or music performance
* Those with more than ten hours of cognitive training

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
N-Back | (CHANGE) up to 16 weeks and after study completion 7 months
  Working Memory Measure in the Visual Domain
Cued Color Word Stroop | (CHANGE) up to 16 weeks and after study completion 7 months
  Cognitive Control, Inhibition
Digit Coding- WAIS IV subtest | (CHANGE) up to 16 weeks and after study completion 7 months
  Simple Processing Speed
Symbol Search- WAIS IV subtest | (CHANGE) up to 16 weeks and after study completion 7 months
  Visual Scanning
Paced Auditory Serial Addition Task (PASAT) | (CHANGE) up to 16 weeks and after study completion 7 months
  Complex processing speed
Rey Auditory Verbal Learning Test | (CHANGE) up to 16 weeks and after study completion 7 months
  Verbal Memory
Delis Kaplan Executive Function Verbal Fluency subtest | (CHANGE) up to 16 weeks and after study completion 7 months
  Category Fluency, Letter Fluency, Category Switching
Trail Making Test | (CHANGE) up to 16 weeks and after study completion 7 months
  Planning and Processing Speed
Finger Tapper Test | (CHANGE) up to 16 weeks and after study completion 7 months
  Motor Speed
Salivary Cortisol | (CHANGE) up to 16 weeks and after study completion 7 months
  Stress Levels
SIgA levels | (CHANGE) up to 16 weeks and after study completion 7 months
  Immune Function
Musical Performance Self-Efficacy | (CHANGE) up to 16 weeks and after study completion 7 months
  Musical Self-Efficacy
General Self-Efficacy | (CHANGE) up to 16 weeks and after study completion 7 months
  General Self-Efficacy
Cognitive Self-Report Questionnaire (25) | (CHANGE) up to 16 weeks and after study completion 7 months
  Mood

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bugos, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No, there is no plan to share individual participant data. We plan on publishing all data collectively.

REFERENCES:
- [Result] Smith GE, Housen P, Yaffe K, Ruff R, Kennison RF, Mahncke HW, Zelinski EM. A cognitive training program based on principles of brain plasticity: results from the Improvement in Memory with Plasticity-based Adaptive Cognitive Training (IMPACT) study. J Am Geriatr Soc. 2009 Apr;57(4):594-603. doi: 10.1111/j.1532-5415.2008.02167.x. Epub 2009 Feb 9. PMID 19220558
- [Result] Duff K, Tometich D, Dennett K. The Modified Telephone Interview for Cognitive Status is More Predictive of Memory Abilities Than the Mini-Mental State Examination. J Geriatr Psychiatry Neurol. 2015 Sep;28(3):193-7. doi: 10.1177/0891988715573532. Epub 2015 Feb 26. PMID 25722349
- [Result] Bugos JA, Perlstein WM, McCrae CS, Brophy TS, Bedenbaugh PH. Individualized piano instruction enhances executive functioning and working memory in older adults. Aging Ment Health. 2007 Jul;11(4):464-71. doi: 10.1080/13607860601086504. PMID 17612811
- [Derived] Bugos JA, Wang Y. Piano Training Enhances Executive Functions and Psychosocial Outcomes in Aging: Results of a Randomized Controlled Trial. J Gerontol B Psychol Sci Soc Sci. 2022 Sep 1;77(9):1625-1636. doi: 10.1093/geronb/gbac021. PMID 35134913